CLINICAL TRIAL: NCT05327959
Title: A.L.P.S. Clavicle Plating System for Clavicle Fracture Fixation Post-Market Follow-up Study (Implants and Instrumentation)
Brief Title: A.L.P.S. Clavicle Plating System PMCF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2020-08T
Record Dates: First submitted 2022-03-10; First posted 2022-04-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Clavicle Fracture; Clavicle Injury
Keywords: clavicle
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): The population target is all subjects suffering clavicle fracture suitable for open reduction and internal fixation by the A.L.P.S. Clavicle Plating System in accordance with the IFU.
  Interventions: Device: Clavicle open reduction and internal fixation

INTERVENTIONS:
Device: Clavicle open reduction and internal fixation — Clavicle open reduction and internal fixation using the A.L.P.S. Clavicle Plating System

SUMMARY:
A commercially available product clinical study which aims to confirm the safety, performance, and clinical benefits to the patient of the ALPS Clavicle Plating system for both the implant itself and the instrumentation used during surgery.

DETAILED DESCRIPTION:
The objectives of this observational, prospective study with optional retrospective enrollment are to confirm safety, performance and clinical benefits of the A.L.P.S Clavicle Plating System and its instrumentation by analysis of fracture healing, functional outcome and adverse events.

The safety of the system will be assessed by monitoring the frequency and incidence of adverse events including re-operations. Relation of the events to implant, instrumentation and/or procedure should be specified.

The performance will be evaluated by assessment of fracture/osteotomy healing and functional outcome of all enrolled study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must have a clavicle fracture requiring surgical intervention and be eligible for fixation by locking plate and screws.
* Unilateral or Bilateral fractures.
* Patient must be capable of understanding the doctor's explanation, following doctor's instruction, is able to and willing to complete the protocol required follow-up.
* Patient must have a signed IRB/EC approved informed consent.

Exclusion Criteria:

* Active infection.
* Patients presenting conditions including blood supply limitations, insufficient quantity or quality of bone.
* Patients with mental or neurologic conditions who are unwilling or incapable of giving proper informed consent, following postoperative care instructions.
* Foreign body sensitivity where material sensitivity is suspected, testing is to be completed prior to implantation of the device.
* Patient is a current alcohol or drug abuser
* Patient is a prisoner
* Patient known to be pregnant or breast feeding
* Likely problems with maintaining follow-up program (e.g. patient with no fixed address, long distance, plans to move during course of study)
* Not expected to survive the duration of the follow-up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with fracture healing | 12 months
  Number of subjects with fracture healing will be assessed through 12 months follow-up. Radiologic fracture healing is defined as: Bridging callus or no visible fracture lines on AP and 15-45° cephalic oblique radiographs.

SECONDARY OUTCOMES:
Frequency and Incidence of Adverse Events (Safety) | 12 months
  Monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.
Range of Motion - Total shoulder motion | 12 months
  Range of Motion (affected and contralateral), Forward elevation (maximum arm-trunk angle), External rotation (arm comfortably at side), External rotation (arm at 90 degrees of abduction), Internal rotation (thumb to back) spinous process, Cross-body adduction (antecubital fossa to opposite acromion (cm)
Clinical efficacy of the device is assessed using the American Shoulder and Elbow Surgeons (ASES) Shoulder Score at 12 months follow-up | 12 months
  The ASES scale is 0-100. 100 is the highest score and indicates the greatest function while 0 is the lowest score.
Euroqol Patient Quality of life measured at 12 months follow-up (EQ-5D-5L) | 12 months
  The EuroQol five dimensions questionnaire (EQ-5D-5L) is a five dimensional self-assessment that is comprised of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These five dimensions can be used to index a subject's health utility on a scale of 0 to 1, where 0 is death and 1 is perfect health. The scoring rule for EQ-5D permits scores less than 0, implying that some health states may be worse than death.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (5):
- United States (4):
  - Cleveland Clinic Florida, Weston, Florida
  - University of Michigan - Michigan Medicine, Ann Arbor, Michigan
  - Slocum Research & Education Foundation, Eugene, Oregon
  - University of Texas San Antonio, San Antonio, Texas
- General Foundation of the University of Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No